CLINICAL TRIAL: NCT05290428
Title: The Accuracy of Host DNA PAX1 and JAM3 Methylation for Cervical Cancer Screening: a Multi-center, Double-blind, Parallel Controlled Clinical Trials
Brief Title: DNA PAX1 and JAM3 Methylation for Cervical Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Other Study IDs: METHY4
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia; DNA Methylation; Cancer Screening; Detection Accuracy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Cervical cytology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective part: This part will enroll at least 120 cases in previously preserved samples.
  Interventions: Diagnostic Test: DNA methylation testing
- Prospective part: This part will enroll at least 339 cases.
  Interventions: Diagnostic Test: DNA methylation testing

INTERVENTIONS:
Diagnostic Test: DNA methylation testing — All cervical cytology samples will be tested for PAX1 and JAM3 methylation

SUMMARY:
Based on the previous study of NCT03961191 and NCT03960879, we performed this trial to further confirm the accuracy of host DNA PAX1 and JAM3 methylation for cervical cancer screening. This study would provide profound basis for the approval of assay kit of DNA methylation in China for cervical screening. Three hospitals, including Peking Union Medical College Hospital, would enroll eligible patients in this study. The cervical cytology of 3 ml will be collected for the detection of DNA PAX1 and JAM3 methylation, and the results will compared with the cervical histological pathology, which is achieved after collection of cervical cytology, by surgeries including loop electrosurgical excision procedure, cervical conization, total hysterectomy and others. The methylation testing would be double-blinded in operators and analysts. The retrospective and prospective parts will enroll at least 120 patients and at least 339 patients, respectively.

ELIGIBILITY:
Inclusion Criteria:

* With uterine cervix intact
* Aged 18 years or older
* With accessible histological results of cervix
* Signed an approved informed consents
* With accessible cervical cytology before harvesting cervical histology

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will accept surgeries harvesting cervical histology.
Sampling Method: Non-Probability Sample
Enrollment: 459 (Estimated)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-09-12 (Estimated); Study Completion 2022-12-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of methylation testing | One week
  Sensitivity of methylation testing of cervical cytology compared with histology
Specificity of methylation testing | One week
  Specificity of methylation testing of cervical cytology compared with histology

SECONDARY OUTCOMES:
Positive predictive value of methylation testing | One week
  Positive predictive value of methylation testing of cervical cytology compared with histology
Negative predictive value of methylation testing | One week
  Negative predictive value of methylation testing of cervical cytology compared with histology

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China